CLINICAL TRIAL: NCT03367572
Title: Netupitant/Palonosetron Hydrochloride and Dexamethasone With or Without Prochlorperazine or Olanzapine in Improving Chemotherapy-Induced Nausea and Vomiting in Patients With Breast Cancer
Brief Title: Treatment of Refractory Nausea and Vomiting in Patients With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester NCORP Research Base (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Luke Peppone, Associate Professor of Surgery and Orthopaedics, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: URCC16070; NCI-2017-00902 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC16070 (Other: University of Rochester NCORP Research Base); URCC-16070 (Other: DCP); R01CA200579 (NIH); UG1CA189961 (NIH)
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; netupitant; Palonosetron; netupitant, palosentron drug combination; Olanzapine; Prochlorperazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (netupitant/palonosetron hydrochloride, dexamethasone (Experimental): Within 1 hour prior to chemotherapy, patients receive netupitant/palonosetron hydrochloride PO on day 1. Within 30 minutes prior to chemotherapy, patients also receive dexamethasone PO on days 1-4. Patients also receive placebo PO with chemotherapy Q8H on days 1-4.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Netupitant/Palonosetron Hydrochloride; Other: Placebo; Other: Quality-of-Life Assessment
- Group II (net/pal hydro, dexa, prochlorperazine, placebo) (Experimental): Patients receive netupitant/palonosetron hydrochloride and dexamethasone as in Group I. Patients also receive prochlorperazine PO Q8H and placebo PO with chemotherapy on days 1-4.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Netupitant/Palonosetron Hydrochloride; Other: Placebo; Drug: Prochlorperazine; Other: Quality-of-Life Assessment
- Group III (net/pal hydro, dexa, olanzapine, placebo) (Experimental): Patients receive netupitant/palonosetron hydrochloride and dexamethasone as in Group I. Patients also receive olanzapine PO and placebo PO Q8H with chemotherapy on days 1-4.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Netupitant/Palonosetron Hydrochloride; Drug: Olanzapine; Other: Placebo; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Netupitant/Palonosetron Hydrochloride — Given PO
  Other Names: Akynzeo
Drug: Olanzapine — Given PO
  Other Names: LY 170053; Zydis; Zyprexa; Zyprexa Zydis
  Arms: Group III (net/pal hydro, dexa, olanzapine, placebo)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
Drug: Prochlorperazine — Given PO
  Other Names: RP 6140; SKF-4657
  Arms: Group II (net/pal hydro, dexa, prochlorperazine, placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies how well netupitant/palonosetron hydrochloride and dexamethasone with prochlorperazine or olanzapine work compared to netupitant/palonosetron hydrochloride and dexamethasone in improving chemotherapy-induced nausea and vomiting in patients with breast cancer. Antiemetic drugs, such as prochlorperazine and olanzapine, may help lessen nausea and vomiting in patients with breast cancer treated with chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if control of nausea at cycle 2 in participants who experienced chemotherapy-induced nausea and vomiting (CINV) at cycle 1 is improved by the addition of either prochlorperazine or olanzapine to the control arm of netupitant, palonosetron and dexamethasone.

SECONDARY OBJECTIVES:

I. To determine if olanzapine is more effective than prochlorperazine in controlling nausea at cycle 2 in participants who experienced CINV at cycle 1 when used in combination with netupitant, palonosetron and dexamethasone.

II. To determine if control of vomiting at cycle 2 in patients who experienced CINV at cycle 1 is improved by the addition of either prochlorperazine or olanzapine to the control arm of netupitant, palonosetron and dexamethasone.

III. To determine if olanzapine is more effective than prochlorperazine in controlling vomiting at cycle 2 in participants who experienced CINV at cycle 1 when used in combination with netupitant, palonosetron and dexamethasone.

TERTIARY OBJECTIVES:

I. To create an empirically-based algorithm predicting nausea from breast cancer chemotherapy regimens that takes into account not only state-of-the-art anti-emetic regimens but also participant factors such as age, race, education, ethnicity, quality of life (QOL), alcohol consumption, susceptibility to nausea, expectancy, anxiety, level of nausea on the day prior to treatment, and prior history of nausea.

II. To compare the effects of the interventions on QOL, as assessed by the Functional Assessment of Cancer Therapy- General (FACT-G), by following the same procedures described under the primary aim and the first secondary aim, using change in the FACT-G scores as the response.

III. To provide preliminary data on the frequency and severity of sleep disturbance, fatigue, anxiety, and dizziness, across treatment conditions.

IV. To provide preliminary data on biological factors (e.g. glutathione [GSH] recycling, genetic markers) that may help identify a subgroup of patients at high risk for development of cancer-related or treatment-related side effects, or response to treatment.

OUTLINE:

PART I: Patients receive 1 cycle of standard of care chemotherapy.

PART II: Patients with a nausea score >= 3 at least once on the diary at cycle 1 chemotherapy are randomized into 1 of 3 groups at cycle 2.

GROUP I: Within 1 hour prior to chemotherapy, patients receive netupitant/palonosetron hydrochloride orally (PO) on day 1. Within 30 minutes prior to chemotherapy, patients also receive dexamethasone PO on days 1-4. Patients also receive placebo PO with chemotherapy every 8 hours (Q8H) on days 1-4.

GROUP II: Patients receive netupitant/palonosetron hydrochloride and dexamethasone as in Group I. Patients also receive prochlorperazine PO Q8H and placebo PO with chemotherapy on days 1-4.

GROUP III: Patients receive netupitant/palonosetron hydrochloride and dexamethasone as in Group I. Patients also receive olanzapine PO and placebo PO Q8H with chemotherapy on days 1-4.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of breast cancer and be chemotherapy naive; NOTE: prior methotrexate for non-cancerous conditions is allowed
* Be scheduled to receive a single-day chemotherapy regimen that contains doxorubicin and/or cyclophosphamide and/or carboplatin. Single-day chemotherapy is defined as only one infusion or injection per cycle. Herceptin (trastuzumab) and other chemotherapy agents will be allowed with any of these regimens
* Be scheduled to receive an antiemetic regimen that does not contain Akynzeo; in addition, the antiemetic regimen must conform with American Society of Clinical Oncology (ASCO) Clinical Practice Guidelines at cycle 1
* Be able to read English
* Have the ability to give written informed consent
* Have Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* NOTE: patients 80 years of age or older must have approval from an oncologist or their designee to participate in this study
* NOTE: patients currently receiving warfarin must have approval from an oncologist or their designee to participate in this study
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, or abstinence) for the duration of the study and have a negative pregnancy test within 10 days prior to the initiation of chemotherapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* CYCLE II PORTION ONLY: Only participants with a nausea score >= 3 at least once on the diary assessment from cycle 1 can be randomized for cycle 2
* CYCLE II PORTION ONLY: Participants must be scheduled to receive the same chemotherapy regimen as received at cycle 1

Exclusion Criteria:

* Have clinical evidence of current or impending bowel obstruction
* Have a known history of central nervous system disease (e.g., brain metastases or a seizure disorder)
* Have dementia
* Have uncontrolled diabetes mellitus or uncontrolled hyperglycemia
* Have severe hepatic impairment, severe renal impairment, or end-stage renal disease as determined by the treating physician
* Have had long term treatment (> 5 days within the past 30 days) with an antipsychotic agent such as risperidone, quetiapine, clozapine, a phenothiazine, or a butyrophenone within 30 days before enrollment or plans for such treatment during the study period; NOTE: participants could have received prochlorperazine and other phenothiazines as antiemetic therapy on a short term basis (i.e., =< 5 days)
* Have a known cardiac arrhythmia, uncontrolled congestive heart failure, or acute myocardial infarction within the previous 6 months
* Be taking benzodiazepines regularly (> 5 days within the past 30 days); pro re nata (PRN) use (=< 5 days) for the short-term relief of the symptoms of anxiety, anxiety associated with depressive symptoms, or as a rescue medication for breakthrough CINV is allowed
* Be taking anticholinergic medications
* Be receiving quinolone antibiotic therapy
* Be taking amifostine (Ethiofos)
* Have a known hypersensitivity to olanzapine or to phenothiazines
* CYCLE II PORTION ONLY: Must not have received Akynzeo at cycle 1
* CYCLE II PORTION ONLY: Must still meet all the exclusion criteria for cycle 1

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1363 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luke Peppone, Principal Investigator — University of Rochester NCORP Research Base
Locations (18):
- United States (18):
  - Hawaii MU NCORP, Honolulu, Hawaii
  - Decatur Memorial Hospital, Decatur, Illinois
  - Gulf South MU-NCORP, New Orleans, Louisiana
  - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Cancer Research Consortium of West Michigan, Grand Rapids, Michigan
  - Health Partners Inc, Minneapolis, Minnesota
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - University of Rochester NCORP Research Base, Rochester, New York
  - Southeast Clinical Oncology Research Program, Winston-Salem, North Carolina
  - Columbus NCORP, Columbus, Ohio
  - Dayton Clinical Oncology Program, Dayton, Ohio
  - Geisinger Cancer Institute NCORP, Danville, Pennsylvania
  - Greenville NCORP, Greenville, South Carolina
  - Upstate Carolina NCORP, Spartanburg, South Carolina
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Gundersen Health System, La Crosse, Wisconsin
  - Aurora NCORP, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1363 subjects were enrolled. CYCLE 1 which is the First Chemotherapy Cycle (excluded 796 [5 registration errors, 41 no four-day home record, 750 did not have average score of 3 or better]) CYCLE 2 which is the Second Chemotherapy Cycle (excluded 250 [subject decided not to continue on cycle 2]). 317 subjects are available for randomization. 310 subjects were actually randomized.
Period: Total Subjects Randomized
Arm/Group | Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone | Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) | Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo)
Started | 92 | 113 | 112
Completed | 91 | 110 | 109
Not Completed | 1 | 3 | 3
Period: Second Chemotherapy Cycle (Cycle 2)
Arm/Group | Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone | Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) | Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo)
Started | 91 | 110 | 109
Completed | 85 | 108 | 100
Not Completed | 6 | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone | Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) | Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo) | Total
Number analyzed (Participants) | 91 | 110 | 109 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (11.3) | 50.0 (11.5) | 50.2 (11.8) | 50.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 110 | 109 | 310
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 5 | 13
  Not Hispanic or Latino | 79 | 102 | 99 | 280
  Unknown or Not Reported | 8 | 4 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 2 | 7 | 6 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 14 | 15 | 38
  White | 75 | 86 | 84 | 245
  More than one race | 2 | 2 | 1 | 5
  Unknown or Not Reported | 3 | 0 | 2 | 5
Marital Status [Count of Participants; unit: Participants]
  Married / Long Term | 66 | 86 | 81 | 233
  Divorced | 8 | 7 | 3 | 18
  Separated | 4 | 2 | 6 | 12
  Single | 10 | 11 | 15 | 36
  Widowed | 3 | 4 | 4 | 11
Education [Count of Participants; unit: Participants]
  College or Grad School | 20 | 27 | 23 | 70
  High School or Less | 71 | 83 | 86 | 240

OUTCOME MEASURES:

1. Primary Outcome: Average Nausea Defined as the Average [ MAXIMUM ] Nausea Rating Across 15 Assessment Points at Cycle 1 and 16 Assessment Points at Cycle 2 (Comparing Prochlorperazine or Olanzapine to Control Arm)
Description: Will be measured on a 7-point scale ("1: not at all nauseated", "4: moderately nauseated", "7: extremely nauseated"). Higher score is a worse outcome. This is averaged over 15 assessment points for Cycle 1 (Day 1 measured at afternoon, evening and night and Days 2 through 4 measured at morning, afternoon, evening and night). This is averaged over 16 assessment points for Cycle 2 (Days 1 through 4 measured at morning, afternoon, evening and night).
Time Frame: Nausea measured at Cycle 1 Chemotherapy (15 time points which is Days 1,2,3,4) and also measured at Cycle 2 Chemotherapy (16 time points which is Days 1,2,3,4)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone | Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) | Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo)
Number analyzed (Participants) | 91 | 110 | 109
units on a scale
  Cycle 1 | 4.51 (0.155) | 4.70 (0.141) | 4.93 (0.141)
  Cycle 2 | 3.22 (0.164) | 2.68 (0.147) | 2.37 (0.152)
Statistical Analysis 1: Comparison: Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone vs Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo); Test type: Superiority; p = 0.008, ANOVA; Mean Difference (Net) = 0.7056
Statistical Analysis 2: Comparison: Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone vs Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo); Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Net) = 1.1486

2. Primary Outcome: Average Nausea Defined as the [AVERAGE] Nausea Rating Across 15 Assessment Points at Cycle 1 and 16 Assessment Points at Cycle 2 (Comparing Prochlorperazine or Olanzapine to Control Arm)
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone | Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) | Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo)
Number analyzed (Participants) | 91 | 110 | 109
units on a scale
  Cycle 1 | 2.40 (0.120) | 2.58 (0.109) | 2.50 (0.109)
  Cycle 2 | 1.90 (0.101) | 1.62 (0.090) | 1.45 (0.093)
Statistical Analysis 1: Comparison: Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone vs Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo); Test type: Superiority; p = 0.010, ANOVA; Mean Difference (Net) = 0.4468
Statistical Analysis 2: Comparison: Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone vs Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo); Test type: Superiority; p = 0.001, ANOVA; Mean Difference (Net) = 0.5632

3. Secondary Outcome: The Secondary Outcome Variable Will be [ MAXIMUM ] Nausea (Measured on a 7-point Scale Anchored by ("1:Not at All Nauseated" and 7:"Extremely Nauseated"). Difference of Average Nausea Between Control and Experimental Arms Will be Calculated and Compared.
Description: Will be measured on a 7-point scale anchored by "1:not at all nauseated" and "7:extremely nauseated". Higher score is a worse outcome. This is averaged over 15 assessment points for Cycle 1 and 16 assessment points for Cycle 2. This will be assessed by estimating the contrast D = (3 - 1) - (2 - 1), where 3 is the Arm 3 mean, 2 is the Arm 2 mean, and 1 is the Control mean.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone | Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) | Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo)
Number analyzed (Participants) | 91 | 110 | 109
units on a scale
  Cycle 1 | 4.51 (0.155) | 4.70 (0.141) | 4.93 (0.141)
  Cycle 2 | 3.22 (0.164) | 2.68 (0.147) | 2.37 (0.152)
Statistical Analysis 1: Comparison: Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) vs Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo); Secondary Aim 1 is to determine if olanzapine is more effective than prochlorperazine in controlling nausea at Cycle 2 in participants who experienced CINV at Cycle 1 when used in combination with netupitant, palonosetron and dexamethasone. This will be assessed by estimating the contrast D = (3 - 1) - (2 - 1), where 3 is the Arm 3 mean, 2 is the Arm 2 mean, and 1 is the Control mean, and testing whether D = 0 versus the one-sided alternative hypothesis that D > 0; Test type: Superiority; p = 0.019, t-test, 2 sided; Mean Difference (Net) = -0.59

4. Secondary Outcome: Vomiting (Yes/No) at Cycle 2 in Participants Who Experienced CINV at Cycle 1.
Description: The response variable will be Any VOMITING (yes/no) after Cycle 2 Chemotherapy, treatment arm as the main factor, and Any Vomiting after Cycle 1 as a covariate. Estimation will be performed using maximum likelihood assuming a binomial distribution and logit link. The same group of contrasts described in the Primary Aim analysis will be estimated and tested, with a significance level of 0.025 to adjust for multiple tests.
Time Frame: Vomiting measured at Cycle 1 Chemotherapy (Yes/No on Days 1,2,3,4) and also measured at Cycle 2 Chemotherapy (Yes/No on Days 1,2,3,4)
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone | Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) | Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo)
Number analyzed (Participants) | 91 | 110 | 109
Participants
  Yes | 7 | 4 | 2
  No | 79 | 103 | 98
  Unknown | 5 | 3 | 9
Statistical Analysis 1: Comparison: Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) vs Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo); Test type: Superiority; p = 0.386, Regression, Logistic — prochlorperazine arm statistics; Odds Ratio (OR) = 1.31, 97.5% CI 2-sided [0.65 to 2.66]
Statistical Analysis 2: Comparison: Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) vs Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo); Test type: Superiority; p = 0.036, Regression, Logistic — olanzapine arm statistics; Odds Ratio (OR) = 0.16, 97.5% CI 2-sided [0.02 to 1.13]

5. Other Pre Specified Outcome: Regimens: Chemotherapy Regimens at Cycle 2
Description: Grouping of Chemotherapy Regimens at Cycle 2
Time Frame: Cycle 2 Chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone | Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) | Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo)
Number analyzed (Participants) | 91 | 110 | 109
Participants
  Anthracycline based | 54 | 68 | 55
  Taxane based | 19 | 22 | 22
  Platinum based | 14 | 16 | 27
  Others | 0 | 2 | 3
  Unknown | 4 | 2 | 2

6. Other Pre Specified Outcome: Emetogenic Potential
Description: Emetogenic Potential: The percentage of risk of vomiting based on given chemotherapy agents. Reference: https://pubmed.ncbi.nlm.nih.gov/38129530/
Time Frame: Cycle 2 Chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone | Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) | Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo)
Number analyzed (Participants) | 91 | 110 | 109
Participants
  High ( >=90 % risk of vomiting ) | 54 | 68 | 55
  Moderate ( 30 - 90 % risk of vomiting ) | 33 | 40 | 52
  Unknown | 4 | 2 | 2

7. Other Pre Specified Outcome: Vomiting at Cycle 1 of Chemotherapy
Description: Record of any vomiting (Yes/No) during Cycle 1 of Chemotherapy on Days 1, 2, 3, 4
Time Frame: Cycle 1 Chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone | Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) | Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo)
Number analyzed (Participants) | 91 | 110 | 109
Participants
  Yes | 12 | 18 | 19
  No | 79 | 92 | 90

8. Other Pre Specified Outcome: Vomiting at Cycle 2 of Chemotherapy
Description: Record of any vomiting (Yes/No) during Cycle 2 of Chemotherapy on Days 1, 2, 3, 4
Time Frame: Cycle 2 Chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone | Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) | Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo)
Number analyzed (Participants) | 91 | 110 | 109
Participants
  Yes | 7 | 4 | 2
  No | 79 | 103 | 98
  Unknown | 5 | 3 | 9

ADVERSE EVENTS:
Time Frame: The time frame for the Adverse Events is within 4 days of when drugs were given at Cycle 2.
Arm/Group | Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone | Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) | Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo)
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/110 | 0/109
Serious Adverse Events (participants affected / at risk) | 1/91 | 3/110 | 3/109
Other Adverse Events (participants affected / at risk) | 10/91 | 19/110 | 14/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone (N=91) | Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) (N=110) | Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo) (N=109)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorders, other specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Netupitant/Palonosetron Hydrochloride, Dexamethasone (N=91) | Group II (Net/Pal Hydro, Dexa, Prochlorperazine, Placebo) (N=110) | Group III (Net/Pal Hydro, Dexa, Olanzapine, Placebo) (N=109)
Headache (Investigations) | 1 (1) | 0 (0) | 0 (0)
Restlessness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 5 (5)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 10 (10) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 4 (4) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Lethargy (General disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Concentration Impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT03367572/Prot_SAP_002.pdf
  • Informed Consent Form (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT03367572/ICF_001.pdf